CLINICAL TRIAL: NCT02853019
Title: Influence of Emotion and Motivation on Behaviour and Neural Activity in Patients With Psychosis
Brief Title: Emotion and Motivation in Patients With Psychosis
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: not enough patients avalaible
Sponsor: University Hospital, Strasbourg, France (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 6152
Record Dates: First submitted 2016-05-23; First posted 2016-08-02 (Estimated); Last update posted 2025-08-19 (Actual); Status verified 2024-08

CONDITIONS: Schizophrenia
Keywords: Emotion; motivation; cognition; schizophrenia
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Healthy volunteers (Sham Comparator): Healthy volunteers
  Interventions: Other: Electroencephalogram; Behavioral: Cognitive tasks; Behavioral: subjective evaluation scales
- Patients with schizophrenia (Experimental): Patients with schizophrenia
  Interventions: Other: Electroencephalogram; Behavioral: Cognitive tasks; Behavioral: subjective evaluation scales

INTERVENTIONS:
Other: Electroencephalogram — electrophysiological measurements (evoked potentials) based on neural activity when visualizing stimuli
Behavioral: Cognitive tasks — - clinical scales and subjective assessments of emotional and motivational stimuli
Behavioral: subjective evaluation scales — - clinical scales and subjective assessments of emotional and motivational stimuli

SUMMARY:
Anhedonia and avolition reflect emotional and motivational disorders, respectively. However, if these disorders play a major role in the symptomatology of schizophrenia, their mechanisms remain poorly understood, and existing treatments are inefficient on these symptoms. The literature suggests that the impairment does not concern emotion or motivation per se, but rather their influence on cognition. This project aims at using recent advances in the fundamental domain to better understand the cognitive and neuronal mechanisms of the patients' alterations, and especially how emotion and motivation influence cognition in schizophrenia.

ELIGIBILITY:
Inclusion Criteria:

* diagnostic and Statistical Manual of Mental Disorders criteria for schizophrenia

Exclusion Criteria:

* addiction problem
* invalidating visual sensory problems
* neurological history
* for the healthy volunteers: psychiatric history

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 41 (Actual)
Dates: Start 2017-02-02 (Actual); Primary Completion 2025-06-01 (Actual); Study Completion 2025-06-01 (Actual)

PRIMARY OUTCOMES:
Change in the amplitude of the CNV (Contingent Negative Variation) as a function of the primer displayed on the screen | During EEG sessions, at experimental session 1 (Day 0) and experimental session 2 (up to Day 120)
  Before each cognitive trial a primer will be displayed, which will be either neutral or convey emotion or motivation. The investigators will check whether this primer affects the subjects preparation by measuring the CNV, which is an evoked potential recorded with electroencephalography, and indexing preparatory effort.

SECONDARY OUTCOMES:
Change in the amplitude of the LPP (Late Positive Potential) as a function of the primer displayed on the screen | During EEG sessions, at experimental session 1 (Day 0) and experimental session 2 (up to Day 120)
  The investigators will check whether primers affect the subjects attention by measuring the LPP, which is an evoked potential recorded with electroencephalography, and indexing sustained attention.

CONTACTS AND LOCATIONS:
Locations (1):
- Unité INSERM 1114, Strasbourg, France

IPD SHARING:
Plan to Share IPD: No